CLINICAL TRIAL: NCT01666145
Title: Advanced Image Guidance for Ablation Probe Placement in Laparoscopic Liver Surgery: A Pilot Study
Brief Title: Advanced Image Guidance Utilized in Liver Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: InnerOptic (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-11-13B
Record Dates: First submitted 2012-05-07; First posted 2012-08-16 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Cancer; Hepatocellular Carcinoma; Hepatoma; Liver Cancer, Adult; Liver Cell Carcinoma, Adult
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraoperative Imaging (Experimental): Laparoscopic microwave ablation surgery utilizing the Advanced Image Guidance system for needle placement.
  Interventions: Device: Advanced Image Guidance

INTERVENTIONS:
Device: Advanced Image Guidance — Patients with hepatocellular carcinoma will be treated through laparoscopic microwave ablation surgery, in which the surgeon will utilize a new guidance system for needle placement.
  Other Names: AIM

SUMMARY:
Advanced Image Guidance for this study was used during laparoscopic microwave ablation surgery to help the surgeon accurately place the ablation needle into the tumor of patients diagnosed with liver cancer.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is diagnosed in over 19,000 Americans annually and responsible for 17,000 deaths. Worldwide, (HCC) is the third leading cause of cancer death. Hepatocellular carcinoma recurs frequently due to its multi-centric nature, which requires repeated treatments and often results in progressively fewer treatment options because of severe underlying liver dysfunction. While surgery offers the best prognosis for such tumors and lesions, only 10-15% of all patients are candidates for removal by surgical means, necessitating the exploration of other treatment options. InnerOptic's AIM Guidance System is designed to alleviate the difficulty in using ultrasound to place a needle. AIM shows the needle and the ultrasound slice in their locations in 3D on a stereo monitor, making the spatial relationship between them obvious. AIM also displays the needle trajectory and where the needle will intersect with the ultrasound image, providing the surgeon with an indication of where the needle will go, if inserted along the needle shaft. AIM can also render an ablation volume guide, providing the surgeon with further confirmation that the needle is placed accurately and providing a volumetric guide regarding the power settings of the ablation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have hepatocellular carcinoma.
* Individuals who are candidates for microwave ablation surgery.

Exclusion Criteria:

* Individuals who do not have hepatocellular carcinoma.
* Individuals who are not a candidate for laparoscopic microwave ablation surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Iannitti, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Health System, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraoperative Imaging
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Imaging
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 63 [47 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Successful Insertion of Ablation Antenna Into Target Lesion
Description: Once the ablation antenna has been placed into the target lesion, the success or failure of the attempt will be confirmed with conventional ultrasound alone, in two planes. If the placement is deemed successful, the surgeon will commence the ablation of the tumor. If the placement is deemed insufficient, the probe will be removed and another placement will be attempted using conventional guidance.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 2 to 3 days.
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Imaging
Number analyzed (Participants) | 14
percentage of participants | 100

2. Secondary Outcome: Percentage of Participants With Significant Ease of Lesion Targeting Using Advanced Image Guidance (AIM)
Description: A subjective grading scale from which the surgeon will provide the relative ease of lesion targeting using Advanced Image Guidance (AIM) and the guidance system; the scale will be numbered 1-5 with one being significantly difficult and five being significantly easy. The percentage of participants with a score of 5 is reported below.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 2 to 3 days.
Measure: Number; unit: percentage of participants
Arm/Group | Intraoperative Imaging
Number analyzed (Participants) | 14
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: To hospital discharge, up to one week
Arm/Group | Intraoperative Imaging
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No